CLINICAL TRIAL: NCT04282382
Title: A Retrospective Analysis of Perioperative Transfusion Management in Children
Brief Title: Intraoperative Transfusion Practice in Children
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Dr. Florian Piekarski, Principle Investigator, Johann Wolfgang Goethe University Hospital
Other Study IDs: KGU_FP_2020_CA5
Record Dates: First submitted 2020-02-17; First posted 2020-02-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Transfusion
Keywords: Transfusion, Pediatric, Patient Blood Management

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to examine factors, impact and outcome on perioperative blood transfusion for pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Operation
* Anaesthesia
* Transfusion (pRBC, plasma or platelets)

Exclusion Criteria:

* No

Ages: 0 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: All pediatric patients being operated an receiving transfusion will be included.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Number of children being transfused intraoperative | 01.04.2018 to 31.10.2019
  Amount of transfused pRBC, plasma, thrombocytes will be evaluated in children undergoing surgery
Documented transfusion indication | 01.04.2018 to 31.10.2019
  Physiologic transfusion triggers will be evaluated (Hb Level, lactate, venous O2 saturation, levels of catecholamines)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesiology, Intensive Care Medicine and Pain Therapy, University Hospital Frankfurt, Goethe University, Frankfurt, North Rhine-Westphalia, Germany